CLINICAL TRIAL: NCT04545320
Title: Effectiveness of Once-a-week High-intensity Interval Training (HIIT) Versus Moderate-intensity Continuous Training (MICT) in Reducing Visceral Fat in Adults With Central Obesity, a Pilot Randomized Controlled Trial.
Brief Title: Effectiveness of High-intensity Interval Training (HIIT) Versus Moderate-intensity Continuous Training (MICT) in Reducing Visceral Fat in Adults With Central Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled in this study due to the COVID-19 pandemic.
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Parco M. Siu, PhD, Associate Professor & Division Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 303005-RF008-CB
Record Dates: First submitted 2020-09-03; First posted 2020-09-11 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Central Obesity
Keywords: Central Obesity; Visceral Fat; HIIT; MICT
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded from the group allocation and the participants will be instructed not to reveal his/her intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care control group (Placebo Comparator): Subjects in the usual care control group will receive a health education program to provide the usual care information. This program will include 3-month biweekly sessions (70 minutes each session, total 6 sessions) for obesity-related health briefing, dietary caloric restriction advice, lifestyle counselling/consultation and stretching exercise.
  Interventions: Behavioral: Usual care control group
- HIIT group (Experimental): A 3-month intervention of HIIT will be given to participants allocated to this group. The once-a-week HIIT will be performed in small groups on treadmills supervised by certified athletic coaches. Subjects will perform brisk walking for four 4-min bouts at 85%-95% maximal heart rate (HRmax) with a 3-min active recovery walk at 50%-70% HRmax between each session. There will be a 5-min warm-up and cool-down in each exercise session. The duration of each exercise session will be 35 minutes. Heart rate will be continuously monitored during training using Polar M300 with OH1 optical heart rate sensor.
  Interventions: Behavioral: HIIT group
- MICT group (Experimental): A 3-month intervention of MICT will be given to participants allocated to this group. The once-a-week MICT will be performed in small groups on treadmills supervised by certified athletic coaches. Subjects will perform mild walking exercise for ~47 minutes at an intensity of 65-75% HRmax. This exercise volume matches the HIIT volume. Heart rate will be continuously monitored during training using Polar M300 with OH1 optical heart rate sensor.
  Interventions: Behavioral: MICT group

INTERVENTIONS:
Behavioral: Usual care control group — Health education
  Arms: Usual care control group
Behavioral: HIIT group — Once-a-week HIIT
  Arms: HIIT group
Behavioral: MICT group — Once-a-week MICT
  Arms: MICT group

SUMMARY:
Obesity is a major risk factor for cardiovascular disease and diabetes as well as all-cause mortality. The prevalence of obesity has continuously increased in most countries and has doubled in over 70 countries since 1980. The World Health Organization (WHO) estimated in 2014 that ~600 million (13%) adults were obese and ~1.9 billion (39%) were overweight worldwide. Notably, United States and China have the highest numbers of obese adults. According to a national survey in China in 2014 conducted among 146,703 Chinese adults aged 20-59, the prevalence of obesity was 13%, central obesity was 25% and overweight was 41%. In Hong Kong, the Behavioural Risk Factor Survey conducted by the Government in 2016 found 39% of adults were classified as overweight or obese, of which 21% were obese. The prevalence of central obesity has also risen steadily since 1999 in America. By 2030 is projected to reach 55.6% in men, 80.0% in women, 47.6% among girls and 38.9% among boys in the United States. Overweight, obesity and central obesity are now already pandemic public health issues causing heavy burden on healthcare system. Nowadays, lifestyle modification interventions still remain as the primary strategy to manage obesity and obesity-related complications, among which exercise is low-cost and effective. Substantial evidences have demonstrated effectiveness of HIIT and MICT in reducing body adiposity and improving body Anthropometry. However, studies have also pointed out "lack of time" is one of the major barriers preventing patients from exercise participation. Therefore, studies have put focus on low-frequency or low-volume exercise in improving health to reduce time commitment and increase exercise adherence. Among substantial evidence, our recent study demonstrated once-a-week HIIT is effectively in improving body composition. The effectiveness of low-frequency exercise in reducing visceral fat has also been explored. However, a recent meta-analysis showed low-frequency exercise is not effective in reducing visceral fat. Notably, the authors pointed out most of studies included in the meta-analysis adopted cycling exercise modality and they suggested walking or running exercise which recruits more body muscles may exert better results. In this study, we propose to adopt walking exercise modality to fill the research gap identified by the meta-analysis. Also, no study has compared the effectiveness of low-frequency HIIT and MICT in reducing visceral fat determined by magnetic resonance imaging (MRI) previously.

Study aim: to examine the effectiveness of once-a-week high-intensity interval training (HIIT) versus moderate-intensity continuous training (MICT) in reducing visceral fat in adults with central obesity

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 - 60,
2. Central obesity, defined as BMI ≥25 (obesity classification adopted by the Hong Kong Government) with waist circumference of ≥90 cm for men and ≥80 cm for women (abdominal obesity according to the International Diabetes Federation's Chinese ethnic-specific criterion),
3. Males and females will be included to enhance generalizability.

Exclusion Criteria:

1. ≥150 minutes moderate-intensity or ≥75 minutes vigorous-intensity exercise weekly,
2. Regular HIIT or MICT (≥1 weekly) in the past 6 months,
3. Medical history of cardiovascular disease, chronic pulmonary or kidney disease, heart failure, cancer, etc.,
4. Somatic conditions that limit exercise participation (e.g., limb loss),
5. Impaired mobility due to chronic diseases (e.g., chronic arthritis/osteoarthritis, neurological, musculoskeletal and autoimmune diseases),
6. Daily smoking and drinking habit,
7. Surgery, therapy or medication for obesity or weight loss in the past 6 months (e.g., gastric bypass, gastric band, sleeve gastrectomy, gastric reduction duodenal switch, and dietitian-prescribed dietary program).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Visceral fat | 3-month follow-up
  The amounts of visceral fat (VAT) at the abdominal region will be assessed by a 1.5-Teala whole-body scanner. A breath-hold localizer scan will be performed prior to the MRI scan. T1-weighted in-phase images will be obtained by fast spoiled gradient-echo sequences during suspended end-expiration. The VAT and between the thoracic diaphragm and the upper broader of the first sacral vertebra will be manually marked on each transverse image to calculate the volume of abdominal VAT.

SECONDARY OUTCOMES:
Subcutaneous fat | 3-month follow-up
  The amounts of subcutaneous fat (SAT) at the abdominal region will be assessed by a 1.5-Teala whole-body scanner. A breath-hold localizer scan will be performed prior to the MRI scan. T1-weighted in-phase images will be obtained by fast spoiled gradient-echo sequences during suspended end-expiration. The SAT between the thoracic diaphragm and the upper broader of the first sacral vertebra will be manually marked on each transverse image to calculate the volume of abdominal SAT.
Body fat mass | 3-month follow-up
  Total body fat mass will be determined using a full body dual-energy X-ray absorptiometry (DXA) scanner (Explorer S/N 91075, Hologic Inc., Waltham, USA). A trained technician who is blinded to the group allocation will perform the tests and analyze the results.
Body fat percentage | 3-month follow-up
  Total body fat percentage will be determined using a full body dual-energy X-ray absorptiometry (DXA) scanner (Explorer S/N 91075, Hologic Inc., Waltham, USA). A trained technician who is blinded to the group allocation will perform the tests and analyze the results.
Body Mass Index | 3-month follow-up
  BMI will be determined by the equation BMI (kg/m2) = bodyweight/height^2. A calibrated electronic balance(UC-321,A&D Weighing, Australia, 150 kg capacity, ± 0.05 kg accuracy) and a stadiometer (Seva 231, Seca, Germany, 205 cm limit, ± 0.05 cm accuracy; ) will be used for the measurements.
Waist Circumference 1 | 3-month follow-up
  Waist circumference will be measured on bare skin midway between the lowest rib and the superior border of the iliac crest using an inelastic measuring tape (Seca 201, Seca, Germany) to the nearest 0.1 cm following the WHO guideline. Measurement will be performed at the end of normal expiration.
Waist Circumference 2 | 3-month follow-up
  Waist circumference will be measured on bare skin following the National Institutes of Health (NIH) guideline method (the superior border of the iliac crest)using an inelastic measuring tape (Seca 201, Seca, Germany) to the nearest 0.1 cm. Measurement will be performed at the end of normal expiration.
Cardiorespiratory fitness | 3-month follow-up
  A maximal exercise test adopting the modified Bruce protocol will be be conducted to determine the maximal oxygen uptake (VO2max) of the subjects. The test will be conducted on a calibrated motor-driven treadmill with continuous metabolic VO2 measurement using a COSMED Quark CPET gas analysis system.
Bone Mineral Density | 3-month follow-up
  Bone mineral density will be simultaneously determined during the DXA scan for total body fat mass.
Lean Mass | 3-month follow-up
  Lean mass will be simultaneously determined during the DXA scan for total body fat mass.
Health-related Quality of Life | 3-month follow-up
  The validated Chinese version 12-item short form survey measures health-related quality of life covering physical functioning, emotional and mental health, bodily pain, general health, vitality, and social functioning. A higher overall score indicates better quality of life.
Adherence | 3-month follow-up
  Class attendance will be analysed to indicate adherence to the interventions.
Adverse Events | 3-month follow-up
  Adverse events will be closely monitored regularly by athletic coaches and research personnel, and by subjects' voluntary reports. Adverse events will be recorded as a secondary outcome.
Medication | 3-month follow-up
  Detailed information (e.g., drug name, type, dose and daily frequency) on the use of dyslipidemic and hypertensive medications will be recorded at baseline. Subjects altering the dosage of medications after consultation with their physician over the study period will also be recorded as a secondary outcome. The lowest recommended dose (LRD) for 7 days will be used for the analysis.
Habitual Physical Activity | 3-month follow-up
  Actigraph activity monitor (wGT3X-BT, Actigraph, USA) worn at the wrist region for 24 h over 7 consecutive days will be used to objectively determine habitual daily physical movement/activities.
Dietary Intake | 3-month follow-up
  Habitual dietary intake will be assessed by 3-day food diary using an electronic scale (KD-400, Tanita, Japan)to determine the daily caloric intake and the relative proportions of macronutrients (carbohydrate, fat, and protein).
Blood pressure | 3-month follow-up
  Blood pressure will be obtained at the same day with blood collection. Subjects will visit our laboratory in the morning after 10 hours of overnight fasting in order to retrain from consuming caffeine, alcohol, and blood pressure drugs at least 10 hours before the assessment. After 10 minutes of seated rest, blood pressure will be measured on the left arm using a sphygmomanometer. Systolic and diastolic blood pressure and mean arterial pressure will be obtained over the brachial artery region with the arm supported at the heart level using an appropriately sized cuff. Three measurements will be taken with a one-minute interval, and the average value will be recorded for analysis.
Hip circumference | 3-month follow-up
  Hip circumference will be be taken on bare skin around the widest portion of the buttocks using an inelastic measuring tape (Seca 201, Seca, Germany) to the nearest 0.1 cm and the tape should be placed parallel to the floor.
Self-report habitual physical activity | 3-month follow-up
  Self-report habitual physical activity will be measured by International Physical Activity Questionnaire (IPAQ). Higher scores indicate higher level of physical activity.
Enjoyment | 3-month follow-up
  Enjoyment towards exercise will be quantitatively measured by the Physical Activity Enjoyment Scale. This Chinese scale has an overall score from 18 to 126. While a higher score indicates higher level of enjoyment towards the exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Fai Parco Siu, PhD, Principal Investigator — Li Ka Shing Faculty of Medicine, The University of Hong Kong
Locations (1):
- Li Ka Shing Faculty of Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data of individual participants that underlie the results reported in this trial, after de-identification including text, tables, figures, and appendices, as well as study protocol and statistical analysis plan, will be shared after 3 months of study publication. Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for the data requests, a data-access agreement needs to be signed.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months after study publication and ending 3 years.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for the data requests, a data-access agreement needs to be signed.